CLINICAL TRIAL: NCT01005771
Title: GF-001001-00 Cream.A Multicentre, Randomised, Double-blind, Parallel, Placebo-controlled Phase II Study to Assess the Efficacy and Safety of 3 Different Doses of GF-001001-00 Cream Versus Placebo Cream Applied 2 Times Daily for 7 Days in the Treatment of Adult Patients With Secondarily-infected Traumatic Lesions
Brief Title: Study to Assess the Efficacy and Safety of GF-001001-00 Cream in Secondarily-Infected Traumatic Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Nuria Albareda, Ferrer Internacional S.A.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-080623-01
Record Dates: First submitted 2009-08-04; First posted 2009-11-02 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Secondarily Infected Traumatic Lesions
Keywords: Secondarily infected traumatic lesions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GF-001001-00 2% (Experimental)
  Interventions: Drug: GF-001001-00
- GF-001001-00 1% (Experimental)
  Interventions: Drug: GF-001001-00
- GF-001001-00 0.25% (Experimental)
  Interventions: Drug: GF-001001-00
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GF-001001-00 — GF-001001-00 2%, 1% and 0.25% twice daily for 7 days
  Arms: GF-001001-00 0.25%; GF-001001-00 1%; GF-001001-00 2%
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, parallel-group, dose-finding study.

DETAILED DESCRIPTION:
200 eligible patients will be included in the double-blind phase (50 in each group, randomised 1:1:1:1 to GF-001001-00 at a concentration of 0.25%, 1% or 2% or placebo).

Randomised patients will apply the study medication as follows depending on their assigned treatment group.

* GF-001001-00 2%, 2 times daily, for 7 days
* GF-001001-00 1%, 2 times daily, for 7 days
* GF-001001-00 0.25%, 2 times daily, for 7 days
* Placebo, 2 times daily, for 7 days

The first application will be done after randomisation at Visit 1 under the guidance of the investigator. Patients will return for control visits: Visit 2 (Day 5) and Visit 3 (Day 7), after randomisation. Patients will return for the Final Visit (Visit 4, Day 14 after initiation of treatment).

Primary objective:

To determine the most effective dose of GF-001001-00 cream for treatment of adult patients with secondarily infected traumatic lesions.

Primary efficacy endpoint:

Clinical response (success or failure) at the Final Visit (Day 14) in the ITTC population.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age.
* Presence of small laceration, sutured wound, abrasion or burn, which has a secondary bacterial infection.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Clinical cure | Day 14

SECONDARY OUTCOMES:
Microbiological cure | Day 14
Adverse events Clinical laboratory parameters Vital signs | Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatologische Praxis, Mahlow, Germany